CLINICAL TRIAL: NCT06374693
Title: Investigating the Tolerability and Feasibility of Transcutaneous Vagus Nerve Stimulation Following Aneurysmal Subarachnoid Haemorrhage
Brief Title: Investigating the Tolerability and Feasibility of tVNS Following aSAH
Acronym: tVNS in aSAH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: STH22772
Record Dates: First submitted 2024-03-25; First posted 2024-04-19 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Subarachnoid Haemorrhage From Cerebral Aneurism Rupture
Keywords: subarachnoid haemorrhage; vagus nerve stimulation; transcutaneous vagus nerve stimulation; aneurysmal subarachnoid haemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stimulation (Experimental): The intervention will take place for 45 minutes twice a day for 5 days after securing the aneurysm
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation
- Sham (Sham Comparator): The placebo group will receive the same intervention, but the device will be in 'sham' mode (i.e. attached to the earlobe).
  Interventions: Device: Sham Transcutaneous Vagus Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Vagus Nerve Stimulation — * Pulse width - 25ms
  * Frequency - device default (20 or 25Hz)
  * Intensity - below pain threshold.
  * Frequency - 45 minutes twice daily. On the basis of similarity to other studies, practicalities on the ward and clinical scenario
  We have chosen a duration of 5 days based on the usual clinical pathway of inpatient management at the Royal Hallamshire Hospital, and have chosen to deliver the treatment twice daily to optimise the dose. This is a pilot study with feasibility outcomes and as such we will be exploring the feasibility of this treatment regimen.
  The Parasym Device will be applied to the left tragus (figure 1) as this is the most common site for tVNS delivery in neurological studies and is associated with few afferents to the heart.
  Arms: Stimulation
Device: Sham Transcutaneous Vagus Nerve Stimulation — The active intervention will be compared to sham tVNS where the vagal nerve stimulator will be attached to the earlobe instead of the tragus, in keeping with evidence that this does not cause vagus nerve stimulation and is in line with sham methods used in other studies. We do not anticipate that patients will have the intervention long enough to become familiar with the common sensations associated with true tVNS intervention. At the end of the intervention period, participants will be asked if they thought they had received true of sham tVNS to understand the blinding ability of the sham.
  Arms: Sham

SUMMARY:
After a subarachnoid haemorrhage, complications are common and increase the overall rate of disability and death from the condition. Despite some advances in preventing, detecting and treating these complications, the rates of complications and associated risks remain high. Further research into ways to reduce complications of subarachnoid haemorrhage.

Transcutaneous vagus nerve stimulation (tVNS) is a technique where a small handheld device is attached to an earpiece which stimulates the nerves to the ear. This is given for short periods and may help improve blood flow and reduce inflammation in the brain. The intervention has been safely used and licensed in seizures, headache and severe depression.

This study will look to see if it is feasible and tolerable to have tVNS twice daily for 5 days after subarachnoid haemorrhage, and whether it can help reduce the risk of complications from subarachnoid haemorrhage.

The participant will be randomly allocated to receive either tVNS or a dummy intervention, known as sham.

The researchers will collect some personal and clinical details such as diagnosis, medications, age, blood test results, as well as some details about the subarachnoid haemorrhage.

The researchers will also complete brief questionnaires with the participant to assess symptoms. They will take measurements of heart rate, pupil response, and brain activity using a cap. The participant will then be randomly allocated to either receive the tVNS or sham intervention.

Next, the research team will apply the earpiece to their ear twice a day for 45 minutes, for a total of 5 days.

At the end of the 5-day study period, the intervention will be complete. The researchers will arrange a follow-up meeting on discharge and at 6 weeks, to assess the participants symptoms and recovery.

Previous studies have shown that tVNS is safe and well tolerated, including a recent review of tVNS studies which evaluated the side effects experienced by 1322 patients receiving tVNS.

The main side effects include localised tingling/numbness/pain/redness around the ear (17%), headaches (3%), dizziness (1%), facial droop (1%), nausea (1%), nasal discharge (2%). Rarely, palpitations or a slow heart rate may occur.

They will continue to receive full medical treatment and observation alongside the study. They are free to withdraw from this study if they find it too demanding on top of their other activities.

DETAILED DESCRIPTION:
The aims of the study will be to conduct a pilot RCT to investigate whether tVNS is a tolerable and feasible treatment for acute aSAH. To understand this the investigators will recruit participants who have recently undergone acute securing procedures follow acute aSAH (coiling or clipping of aneurysm) to a 5 day programme of intervention (active tVNS vs sham) and collect outcome data (primary and secondary as per outcomes section). The investigators will evaluate whether pre-defined success criteria are achieved for tolerability and feasibility and explore signals of effect on clinical outcome measures and mechanistic measures. Non-invasive vagal nerve stimulation has not been studied in the acute period following aSAH outside of the remit of reducing headache. This should offer critical insights as to whether this intervention has potential to take forward to a larger phase 2/3 clinical study.

This is a single centre, pilot, randomised controlled trial. 30 participants who have suffered an aneurysmal subarachnoid haemorrhage and had their aneurysm secured (coiled or clipped successfully).

The intervention will take place for 45 minutes twice a day for 5 days after securing the aneurysm. The placebo group will receive the same intervention, but the device will be in 'sham' mode (i.e. attached to the earlobe).

It is not known whether tVNS is tolerable, and feasible in aSAH, but standard device settings will be used in accordance with a majority of other studies. Similarly, the optimal therapeutic duration is not known - 45 minutes twice a day is a similar usage to other studies. A 5-day course has been chosen because it covers the highest risk period for DCI and is feasible for the research team to deliver.

This is a single centre pilot, single blind, randomised, placebo - controlled study.

This has been chosen as it will demonstrate feasibility and tolerability, whilst providing early data to indicate whether tVNS may provide benefit in this setting, supporting the development of a larger RCT to establish whether it is a statistically significant benefit.

Patients may be able to tell the different between an activated device and sham (where the device is applied to the earlobe instead of the tragus). However, they will not experience both settings, and the investigators will make no clear distinction of exactly what they should feel.

A sample size of at least 30 has been chosen based on the number or participants required for the purposes of a feasibility assessment.9 It is also a practically feasible number of participants to recruit based on annual admission numbers of patients to the RHH (Royal Hallamshire Hospital, Sheffield) and the timeframe of the recruitment period.

Potential participants with aSAH will be identified on admission to neurosurgery at RHH and approached about the study by the clinical treating team on the basis of convenience sampling. If they are interested in the study, they will be provided with an information sheet again and the opportunity to discuss the study with a member of the research team. If they are willing to take part in the study written informed consent will be obtained, after a screening consent support tool is used to ensure the patient had adequate comprehension.

Capacity to consent to the study would be determined by the treating clinical team and confirmed by the research team according to the principles of the mental capacity act (MCA, 2005). Where the patient lacks capacity to consent (including sedated/intubate patients), a personal or nominated consultee can provide advice on what they feel the patients' wishes would be if they had capacity. The treating clinical team would introduce the study to the consultee and an information leaflet given to them. The consultee would then have the option to sign a consent form if they believed the patient would agree to participate. In accordance with the MCA 2005, ongoing consent or assent would be sought from the individual or consultee at each study visit, before any research activity at the that visit is undertaken. Consultees may advise at any point that they believe the person's wishes about participation have changed and they should therefore be withdrawn from the study. Agitated patients will not receive the intervention if they are unable to tolerate it.

The investigators are using tVNS settings that are widely used in other neurological conditions (epilepsy, migraine)14. These include:

* Pulse width - 25ms
* Frequency - device default (20 or 25Hz)
* Intensity - below pain threshold.
* Frequency - 45 minutes twice daily. On the basis of similarity to other studies, practicalities on the ward and clinical scenario

The investigators have chosen a duration of 5 days based on the usual clinical pathway of inpatient management at the Royal Hallamshire Hospital, and have chosen to deliver the treatment twice daily to optimise the dose. This is a pilot study with feasibility outcomes and as such the investigators will be exploring the feasibility of this treatment regimen.

The Parasym Device will be applied to the left tragus (figure 1) as this is the most common site for tVNS delivery in neurological studies and is associated with few afferents to the heart.

The intervention is aimed at supplementing routine clinical care, and as such, the doses of tVNS can be interrupted for care activities (therapy sessions, examinations, assessments etc) and resume afterwards. The overall minute duration will aim to remain 45 minutes twice daily.

The active intervention will be compared to sham tVNS where the vagal nerve stimulator will be attached to the earlobe instead of the tragus, in keeping with evidence that this does not cause vagus nerve stimulation and is in line with sham methods used in other studies. The investigators do not anticipate that patients will have the intervention long enough to become familiar with the common sensations associated with true tVNS intervention. At the end of the intervention period, participants will be asked if they thought they had received true of sham tVNS to understand the blinding ability of the sham.

The investigators will use the FNIRS Lumo ecosystem (Gower labs) to assess cerebral blood flow in the frontal lobes. The investigators will complete a protocol where 6 optodes are placed bilaterally over the frontal and prefrontal cortices. The investigators will complete and record resting state signals of oxyhaemoglobin and deoxyhaemoglobin for 5 minutes while patients are laid in bed with their eyes closed (or wearing an eye patch). Following the 5-minute rest phase, vagal nerve stimulation or sham stimulation will start depending on the participants randomisation and signal acquisition will continue for 5 minutes. After this time, the stimulation will cease and a further 5 minutes of resting signal acquisition will be completed. The data acquired during this protocol will undergo processing (adjustment for background and physiological noise) and data analysis using recommended software (Homer 2/3). Data analysis will look to compare signal acquisition between resting and stimulation states and will evaluate any lasting effects of stimulation following termination. The investigators will perform this on the first and last day of the intervention, before and after stimulation respectively.

The investigators will be using Reflex Pupillometry to measure pupillograms in response to a light stimulus during an intervention session for all participants. This will be done at a different time to the Lumo FNIRS assessment. Recording of the pupillary response will follow the following protocol; 3 baseline measures taken 1 minute apart prior to stimulation will represent baseline pupillograms (which will be averaged). Following this, stimulation (active or sham) will start and 3 times pupillograms will be measured at 1 minute intervals following initiation. After completion of the treatment session, 3 further pupillograms separated by 1-minute intervals will be measured - that will constitute the recovery phase.

Enrolled participants will be issued with a study number and randomised 2:1 (SealedEnvelope Ltd) stratified according to age (<65 and ≥ 65 years). They will then receive either active tVNS stimulation (tragus) or sham (earlobe), twice daily for 45 minutes per session for 5 days. The investigators do not anticipate discharges from hospital earlier than 5 days as this is not routine practice in the neurosurgical unit.

Primary outcome measures of tolerability and feasibility will be collected daily by researchers delivering the intervention, and secondary outcome measures will be collected at the end of intervention or on hospital discharge as detailed in figure 2.

Following discharge from hospital participants will return for follow up clinic assessment at 4 weeks where questionnaire measures of functional recovery and adverse event reporting will be undertaken. After this the participants involvement in the study will be complete.

The analyses will be undertaken on statistical software (PRISM) and will compare the two groups. Rates of complications and outcomes will be reported descriptively. Data integrity will be checked by two researchers and inputted contemporaneously. Each researcher will be trained in outcome measures prior to study initiation.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Admitted to STH (Sheffield Teaching Hospital) neurosurgery department
* Confirmed aneurysmal SAH on vascular imaging
* Within 5 days of 'Securing' aneurysm (i.e., successfully coiled or surgically following rupture)

Exclusion Criteria:

* Current or prior use of a vagus nerve stimulation
* Symptomatic bradycardia or PPM insertion
* Complete heart block
* Implantation of any other electrical stimulator (e.g. DBS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Monitor tolerability for tVNS | 4 weeks
  Symptom severity scores of mild or moderate in less than 1/3 of participants able to report symptoms
Assess study feasibility | 24 months
  recruit >1 patient per month of recruitment, and >80% of recruited patients completing primary outcome measures

SECONDARY OUTCOMES:
Monitor safety criteria for tVNS | 4 weeks
  No SAEs reported to tVNS, and Unexpected AEs in less than 1/3 of participants
Rates of delayed cerebral ischaemia (DCI) | 4 weeks
  Clinical or radiological DCI
Inpatient mortality | 4 weeks
  Inpatient mortality
Length of inpatient stay | From the date of admission to the date of discharge from hospital up to 100 months
  Days
Rates of inpatient complications | From the date of admission to the date of discharge from hospital up to 100 months
  clinically relevant seizures, hyponatraemia, rebleeding, hydrocephalus
Modified rankin score | 4 weeks
  disability score (Score 0-6)
Barthel Index | 4 weeks
  disability score (0-100)
Inflammatory markers | Baseline and end of intervention (day 5)
  Concentration of IL-1beta, IL-6, IL-10, TNF-alpha
Headache scores | 4 weeks
  Likert scale (1 none to 5 severe)
Cerebral functional near-infrared spectroscopy | Baseline and 5 days
  Measure of cerebral cortical blood flow and activation (g/dl oxy and de-oxyhaemoglobin)
Heart rate variability | Baseline and 5 days
  5 minute recording of continuous beat to beat heart rate before and after stimulation with VNS (SDNN)
Pupillary light reactivity | Baseline and 5 days
  Pupillary response to a standardised light stimulus (constriction speed, m/s)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ali Ali, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust; Professor Arshad Majid, Study Director — University of Sheffield
Locations (1):
- University of Sheffield, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2023-12-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT06374693/Prot_000.pdf